CLINICAL TRIAL: NCT03042572
Title: Allogeneic Mesenchymal Stromal Cells for Angiogenesis and Neovascularization in No-option Ischemic Limbs; A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Allogeneic Mesenchymal Stromal Cells for Angiogenesis and Neovascularization in No-option Ischemic Limbs
Acronym: SAIL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Martin Teraa, MD, PhD (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Martin Teraa, MD, PhD, Surgical Resident & Postdoc Physician, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL59038.000.16
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Diseases; Vascular Diseases
Keywords: Critical Limb Ischemia (CLI); Severe Limb Ischemia (SLI); Peripheral Artery Disease (PAD); Peripheral Artery Occlusive Disease (PAOD); Cardiovascular disease; Mesenchymal stromal cell (MSC); Mesenchymal stem cell (MSC)
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Vascular Diseases; Chronic Limb-Threatening Ischemia; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic Mesenchymal Stromal Cell (Experimental): Intramuscular Allogeneic Bone marrow-derived Mesenchymal Stromal Cell Injection
  Interventions: Drug: Allogeneic Mesenchymal Stromal Cell
- Placebo (Placebo Comparator): Intramuscular placebo injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Allogeneic Mesenchymal Stromal Cell — Intramuscular allogeneic BM-MSC injection: MSCs will be extracted from BM of healthy volunteers, expanded with human platelet lysate, and stored. Patients will receive intramuscular allogeneic BM-MSC injections at 30 sites in the lower leg of the ischemic limb. Blinded syringes are provided and cell suspensions will be injected intramuscularly by an experienced operator into multiple sites (30 sites, 1-1.5cm in depth, volume of 1.0mL containing 5*10^6 MSC per site; total 150*10^6 BM-MSCs) in the ischemic lower extremity. Injections will be performed under IV analgesia (fentanyl) and sedation (midazolam) if necessary.
  Other Names: Allogeneic bone marrow-derived mesenchymal stromal cells; Allogeneic bone marrow-derived mesenchymal stem cells; Allogeneic BM-MSC
  Arms: Allogeneic Mesenchymal Stromal Cell
Other: Placebo — Intramuscular placebo injections. Patients will receive intramuscular placebo injections at 30 prespecified sites in the lower leg of the ischemic limb. Blinded syringes are provided and will be injected intramuscularly by an experienced operator into multiple sites (30 sites, 1-1.5cm in depth, volume of 1.0mL placebo per site) in the ischemic lower extremity. Injections will be performed under IV analgesia (fentanyl) and sedation (midazolam) if necessary.
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate whether intramuscular administration of allogeneic mesenchymal stromal cells (MSC) is safe and potentially effective, assessed as a composite outcome of mortality, limb status, clinical status (Rutherford classification) and pain score (visual analogue scale), in patients with no-option severe limb ischemia (SLI).

The investigators will conduct a double-blind, placebo-controlled randomized clinical trial to investigate the effect of allogeneic bone marrow(BM)-derived MSC in patients with SLI, who are not eligible for conventional surgical or endovascular therapies. The investigators intend to include 60 patients, who will be randomized to undergo 30 intramuscular injections with either BM-MSC (30 injection sites with 5*10^6 MSCs each) or placebo in the lower leg of the ischemic extremity. Primary outcome i.e. therapy success, a composite outcome considering mortality, limb status, clinical status (Rutherford classification) and changes in pain score, will be assessed at six months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Severe Peripheral Artery Disease (PAD; Fontaine class III and / or IV):

  * Fontaine III (Rutherford 4): persistent, recurring rest pain requiring analgesia
  * Fontaine IV (Rutherford 5): non-healing ulcers present for > 4 weeks without evidence of improvement in response to conventional therapies
* Ankle brachial index < 0.6 or unreliable (non-compressible or not in proportion to the Fontaine classification)
* Not eligible for surgical or endovascular revascularization
* Written informed consent.

Exclusion Criteria:

* History of neoplasm or malignancy in the past 10 years
* Serious known concomitant disease with life expectancy of less than one year
* Rutherford 6 in which amputation on the short term (within 1-2 weeks) is inevitable
* Pregnancy or unwillingness to use adequate contraception during study
* Uncontrolled acute or chronic infection with systemic symptoms
* Follow-up impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Therapy Success | 6 months
  Composite outcome measure considering mortality, limb status, clinical classification and changes in pain score. To be a "success" a subject must: A, be alive; B, be without a major amputation on the index limb; C, have not worsened in Rutherford classification or visual analog pain scale; and D, have improved in either Rutherford classification or visual analog pain scale. Subjects not meeting all of the criteria are classified as failures.

SECONDARY OUTCOMES:
Major amputation | 2, 6, 12, 24, and 60 months
  Amputation sited proximal from the ankle joint
Minor amputation | 2, 6, 12, 24, and 60 months
  Amputation sited distal from the ankle joint
Therapy Success | 2, 6, 12, 24, and 60 months
  Composite outcome measure considering mortality, limb status, clinical classification and changes in pain score. To be a "success" a subject must: A, be alive; B, be without a major amputation on the index limb; C, have not worsened in Rutherford classification or visual analog pain scale; and D, have improved in either Rutherford classification or visual analog pain scale. Subjects not meeting all of the criteria are classified as failures.
Mortality | 2, 6, 12, 24, and 60 months
  Mortality
Ulcer healing | 2 and 6 months
  Changes in the number and extent of leg ulcers,
Changes in pain | 2, 6, 12, 24, and 60 months
  Resolution of rest pain and alteration in visual analogue pain (VAS) score
Pain-free walking distance | 2 and 6 months
  Changes in pain free walking distance (treadmill at 3 km/h without incline)
Ankle-brachial index (ABI) | 2 and 6 months
  Alterations in ankle-brachial index (ABI)
Toe-brachial index (TBI) | 2 and 6 months
  Alterations in toe-brachial index (TBI)
Quality of life based on EuroQol 5D (EQ5D) questionnaire scores | 2, 6, 12, 24, and 60 months
  Alterations in quality of life assessed using EuroQoL 5D quality of life questionnaire
Quality of life based on Short Form 36 (SF36) questionnaire scores | 2, 6, 12, 24, and 60 months
  Alterations in quality of life assessed using Short Form 36 quality of life questionnaire
Clinical status according to Fontaine classification | 2, 6, 12, 24, and 60 months
  Alterations clinical status according to Fontaine classification
Clinical status according to Rutherford classification | 2, 6, 12, 24, and 60 months
  Alterations clinical status according to Rutherford classification

OTHER OUTCOMES:
Correlation of in-vitro angiogenic assay (Boyden chamber migration assays to test migration towards a platelet derived growth factor gradient) of donor MSC with clinical effect | 6 months
  The investigators will use Boyden chamber migration assays to test migration towards a platelet derived growth factor gradient in order to test angiogenic capacity of the batches of donor Mesenchymal Stromal Cells (MSC) and correlate these with the primary and secondary outcomes (et al. Mol Ther. 2014).
Correlation of in-vitro angiogenic assay (Endothelial repair assay using a scratch wound assay using MSC-derived conditioned medium) of donor MSC with clinical effect | 6 months
  The investigators will use endothelial repair assays using a scratch wound assay with MSC-derived conditioned medium to test angiogenic capacity of the batches of donor Mesenchymal Stromal Cells (MSC) and correlate these with the primary and secondary outcomes (see Gremmels et al. Mol Ther. 2014).
Correlation of in-vitro angiogenic assay (Matrigel tubule forming assay) of donor MSC with clinical effect | 6 months
  The investigators will use matrigel tubule forming assays using MSC-derived conditioned medium to test angiogenic capacity of the batches of donor Mesenchymal Stromal Cells (MSC) and correlate these with the primary and secondary outcomes (see Gremmels et al. Mol Ther. 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne C Verhaar, MD, PhD, Principal Investigator — UMC Utrecht; Gert Jan de Borst, MD, PhD, Study Chair — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Study outcomes will be published in international peer-reviewed journals and individual participant data (IPD) will become available on request.

REFERENCES:
- [Background] Teraa M, Sprengers RW, Schutgens RE, Slaper-Cortenbach IC, van der Graaf Y, Algra A, van der Tweel I, Doevendans PA, Mali WP, Moll FL, Verhaar MC. Effect of repetitive intra-arterial infusion of bone marrow mononuclear cells in patients with no-option limb ischemia: the randomized, double-blind, placebo-controlled Rejuvenating Endothelial Progenitor Cells via Transcutaneous Intra-arterial Supplementation (JUVENTAS) trial. Circulation. 2015 Mar 10;131(10):851-60. doi: 10.1161/CIRCULATIONAHA.114.012913. Epub 2015 Jan 7. PMID 25567765
- [Background] Peeters Weem SM, Teraa M, de Borst GJ, Verhaar MC, Moll FL. Bone Marrow derived Cell Therapy in Critical Limb Ischemia: A Meta-analysis of Randomized Placebo Controlled Trials. Eur J Vasc Endovasc Surg. 2015 Dec;50(6):775-83. doi: 10.1016/j.ejvs.2015.08.018. Epub 2015 Oct 12. PMID 26460286
- [Background] Teraa M, Sprengers RW, van der Graaf Y, Peters CE, Moll FL, Verhaar MC. Autologous bone marrow-derived cell therapy in patients with critical limb ischemia: a meta-analysis of randomized controlled clinical trials. Ann Surg. 2013 Dec;258(6):922-9. doi: 10.1097/SLA.0b013e3182854cf1. PMID 23426345
- [Background] Spreen MI, Gremmels H, Teraa M, Sprengers RW, Verhaar MC, Statius van Eps RG, de Vries JP, Mali WP, van Overhagen H; PADI and JUVENTAS Study Groups. Diabetes Is Associated With Decreased Limb Survival in Patients With Critical Limb Ischemia: Pooled Data From Two Randomized Controlled Trials. Diabetes Care. 2016 Nov;39(11):2058-2064. doi: 10.2337/dc16-0850. Epub 2016 Sep 9. PMID 27612499
- [Background] Teraa M, Conte MS, Moll FL, Verhaar MC. Critical Limb Ischemia: Current Trends and Future Directions. J Am Heart Assoc. 2016 Feb 23;5(2):e002938. doi: 10.1161/JAHA.115.002938. No abstract available. PMID 26908409
- [Background] Peeters Weem SM, Teraa M, den Ruijter HM, de Borst GJ, Verhaar MC, Moll FL. Quality of Life After Treatment with Autologous Bone Marrow Derived Cells in No Option Severe Limb Ischemia. Eur J Vasc Endovasc Surg. 2016 Jan;51(1):83-9. doi: 10.1016/j.ejvs.2015.09.010. Epub 2015 Oct 26. PMID 26511056
- [Background] Teraa M, Schutgens RE, Sprengers RW, Slaper-Cortenbach I, Moll FL, Verhaar MC; Juventas Study Group. Core diameter of bone marrow aspiration devices influences cell density of bone marrow aspirate in patients with severe peripheral artery disease. Cytotherapy. 2015 Dec;17(12):1807-12. doi: 10.1016/j.jcyt.2015.08.004. Epub 2015 Sep 28. PMID 26428987
- [Background] Wisman PP, Teraa M, de Borst GJ, Verhaar MC, Roest M, Moll FL. Baseline Platelet Activation and Reactivity in Patients with Critical Limb Ischemia. PLoS One. 2015 Jul 6;10(7):e0131356. doi: 10.1371/journal.pone.0131356. eCollection 2015. PMID 26148006
- [Background] Gremmels H, Teraa M, Quax PH, den Ouden K, Fledderus JO, Verhaar MC. Neovascularization capacity of mesenchymal stromal cells from critical limb ischemia patients is equivalent to healthy controls. Mol Ther. 2014 Nov;22(11):1960-70. doi: 10.1038/mt.2014.161. Epub 2014 Sep 1. PMID 25174586
- [Background] Gremmels H, Fledderus JO, Teraa M, Verhaar MC. Mesenchymal stromal cells for the treatment of critical limb ischemia: context and perspective. Stem Cell Res Ther. 2013;4(6):140. doi: 10.1186/scrt351. PMID 24246031
- [Background] Teraa M, Fledderus JO, Rozbeh RI, Leguit RJ, Verhaar MC; Juventas Study Groupdagger. Bone marrow microvascular and neuropathic alterations in patients with critical limb ischemia. Circ Res. 2014 Jan 17;114(2):311-4. doi: 10.1161/CIRCRESAHA.114.302791. Epub 2013 Nov 11. PMID 24218170
- [Background] Niemansburg SL, Teraa M, Hesam H, van Delden JJ, Verhaar MC, Bredenoord AL. Stem cell trials for cardiovascular medicine: ethical rationale. Tissue Eng Part A. 2014 Oct;20(19-20):2567-74. doi: 10.1089/ten.TEA.2013.0332. Epub 2013 Dec 11. PMID 24164351
- [Background] Westerweel PE, Teraa M, Rafii S, Jaspers JE, White IA, Hooper AT, Doevendans PA, Verhaar MC. Impaired endothelial progenitor cell mobilization and dysfunctional bone marrow stroma in diabetes mellitus. PLoS One. 2013;8(3):e60357. doi: 10.1371/journal.pone.0060357. Epub 2013 Mar 28. PMID 23555959
- [Background] Teraa M, Sprengers RW, Westerweel PE, Gremmels H, Goumans MJ, Teerlink T, Moll FL, Verhaar MC; JUVENTAS study group. Bone marrow alterations and lower endothelial progenitor cell numbers in critical limb ischemia patients. PLoS One. 2013;8(1):e55592. doi: 10.1371/journal.pone.0055592. Epub 2013 Jan 31. PMID 23383236
- [Background] Setacci C, de Donato G, Teraa M, Moll FL, Ricco JB, Becker F, Robert-Ebadi H, Cao P, Eckstein HH, De Rango P, Diehm N, Schmidli J, Dick F, Davies AH, Lepantalo M, Apelqvist J. Chapter IV: Treatment of critical limb ischaemia. Eur J Vasc Endovasc Surg. 2011 Dec;42 Suppl 2:S43-59. doi: 10.1016/S1078-5884(11)60014-2. PMID 22172473
- [Background] Sprengers RW, Teraa M, Moll FL, de Wit GA, van der Graaf Y, Verhaar MC; JUVENTAS Study Group; SMART Study Group. Quality of life in patients with no-option critical limb ischemia underlines the need for new effective treatment. J Vasc Surg. 2010 Oct;52(4):843-9, 849.e1. doi: 10.1016/j.jvs.2010.04.057. PMID 20598482
- [Background] Sprengers RW, Moll FL, Teraa M, Verhaar MC; JUVENTAS Study Group. Rationale and design of the JUVENTAS trial for repeated intra-arterial infusion of autologous bone marrow-derived mononuclear cells in patients with critical limb ischemia. J Vasc Surg. 2010 Jun;51(6):1564-8. doi: 10.1016/j.jvs.2010.02.020. PMID 20488328
- [Derived] Wijnand JGJ, Teraa M, Gremmels H, van Rhijn-Brouwer FCC, de Borst GJ, Verhaar MC; SAIL Study Group. Rationale and design of the SAIL trial for intramuscular injection of allogeneic mesenchymal stromal cells in no-option critical limb ischemia. J Vasc Surg. 2018 Feb;67(2):656-661. doi: 10.1016/j.jvs.2017.09.026. Epub 2017 Dec 11. PMID 29242062